CLINICAL TRIAL: NCT03249584
Title: OsteoCool Tumor Ablation Post-Market Study (OPuS One)
Brief Title: OsteoCool Tumor Ablation Post-Market Study
Acronym: OPuS One
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT16075
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Metastasis Spine; Metastasis to Bone

STUDY DESIGN:
Intervention Model Description: Enrollment/Baseline visit, OsteoCool procedure visit and 5 post-procedure visits (3 days, 1 week, 1-, 3-, and 6-month clinic visits) and a final post-procedure study visit (12 months) for a total of 8 study related visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- OsteoCool™ RF Ablation (Other): Subjects will undergo a single OsteoCool™ RF Ablation procedure.
  Interventions: Device: OsteoCool™ RF Ablation

INTERVENTIONS:
Device: OsteoCool™ RF Ablation — The OsteoCool™ RF Ablation system is indicated in the United States (US), Europe (EUR) and Canada (CAN) for patients with metastatic malignant lesions in a vertebral body, painful metastatic lesions involving bone (in the US, patients with metastatic lesions involving the bone must have failed or were not candidates for standard therapy) and benign bone tumors such as osteoid osteomas.

SUMMARY:
This study evaluates the effectiveness of the Medtronic OsteoCool™ RF Ablation System.

DETAILED DESCRIPTION:
The OsteoCool™ RF Ablation system has 510k regulatory clearance in the United States, Conformité Européene (CE) mark in Europe, and Health Canada Licence in Canada. The goal of this study is to collect real-world outcomes among a cohort of patients in the US, EUR and CAN with metastatic malignant lesions in a vertebral body, painful metastatic lesions involving bone (in the US, patients with metastatic lesions involving the bone must have failed or were not candidates for standard therapy), and benign bone tumors such as osteoid osteoma who receive treatment with the OsteoCool™ RF Ablation system. Additionally, the study will collect device, procedure and/or therapy related adverse events and device deficiencies. Lastly, subject outcomes (such as pain relief, quality of life, and function) will be evaluated using validated assessment measures.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for OsteoCool RF ablation per the labeled indication applicable in their respective country/region
2. A. Metastatic lesions targeted for treatment must be located in the thoracic and/or lumbar vertebral body(ies), periacetabulum, iliac crest, and/or sacrum OR benign bone tumors - no restrictions on location of lesion
3. Report worst pain score ≥4/10 at the target treatment site within the past 24 hours
4. Localized pain resulting from no more than two sites total of metastatic disease
5. Have Karnofsky score ≥40 at enrollment (not applicable for subjects with benign bone tumors)
6. Willing and able to provide a signed and dated informed consent, comply with the study plan, follow up visits and phone calls
7. At least 18 years old at the time of informed consent

Exclusion Criteria:

1. A. Implanted with heart pacemaker or other implanted electronic device (Europe and Canada only)
2. Use of OsteoCool in vertebral body levels C1-C7
3. Multiple myeloma, solitary plasmacytoma, or primary malignant lesions in the index vertebra or bone
4. Active or incompletely treated local infection at the planned treatment site(s) and/or systemic infection
5. Planned treatment site(s) accompanied by objective evidence of secondary radiculopathy or neurologic compromise
6. Planned treatment site(s) associated with spinal cord compression or canal compromise requiring decompression
7. Fractures due to prostatic cancer or other osteoblastic metastases to the spine. Metastatic lesions originating in the prostate that are osteolytic or mixed origin are eligible for the study
8. Pregnant, breastfeeding, or plan to become pregnant during the study duration
9. Concurrent participation in another clinical study that may add additional safety risks and/or confound study results*
10. Any condition that would interfere with the subject's ability to comply with study instructions or might confound the study interpretation

    * Subjects in concurrent studies can only be enrolled with permission from Medtronic. Please contact Medtronic's study manager to determine if the subject can be enrolled in both studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Bagla, MD, Principal Investigator — Vascular Institute of Virginia
Locations (16):
- United States (12):
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Saint Jude Medical Center, Fullerton, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northside Hospital, Cumming, Georgia
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Renown Regional Medical Center, Reno, Nevada
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas (UT) Southwestern Medical Center, Dallas, Texas
  - Vascular Institute of Virginia, Woodbridge, Virginia
- Sunnybrook Health Science Centre, Toronto, Canada
- Hôpitaux Universitaires de Strasbourg - Nouvel Hôpital Civil, Strasbourg, France
- Universitätsklinikum Leipzig AöR, Leipzig, Germany
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levy J, Hopkins T, Morris J, Tran ND, David E, Massari F, Farid H, Vogel A, O'Connell WG, Sunenshine P, Dixon R, Gangi A, von der Hoh N, Bagla S. Radiofrequency Ablation for the Palliative Treatment of Bone Metastases: Outcomes from the Multicenter OsteoCool Tumor Ablation Post-Market Study (OPuS One Study) in 100 Patients. J Vasc Interv Radiol. 2020 Nov;31(11):1745-1752. doi: 10.1016/j.jvir.2020.07.014. PMID 33129427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the time of the primary objective assessment (Apr 2019), 106 subjects were enrolled. Enrollment ended Feb 2020 with 218 total subjects which allowed for assessment of secondary objective and long-term effectiveness and safety.
Pre-assignment Details: 12 of 218 subjects exited prior to RF Ablation (RFA) due to failing in/exclusion criteria, withdrawal of consent, etc. 206 total subjects underwent a single OsteoCool™ RFA procedure. For effectiveness, subjects were separated into 2 study Groups (Thoracic/Lumbar and Periacetabulum/Iliac Crest/Sacrum) based on the location of each subject's ablation(s); subjects were combined for safety.
Groups:
- OsteoCool™ RF Ablation in Thoracic/Lumbar Spine: Subjects underwent a single OsteoCool™ RF Ablation procedure. All ablations were in the Thoracic/Lumbar Spine.
- OsteoCool™ RF Ablation in Periacetabulum/Iliac Crest/Sacrum: Subjects underwent a single OsteoCool™ RF Ablation procedure. At least one ablation was in the Periacetabulum/Iliac Crest/Sacrum. Some subjects also had RF Ablation in the Thoracic/Lumbar in the same procedure.
Period: Overall Study
Arm/Group | OsteoCool™ RF Ablation in Thoracic/Lumbar Spine | OsteoCool™ RF Ablation in Periacetabulum/Iliac Crest/Sacrum
Started (Subjects who received RF Ablation) | 184 | 22
Month 3 | 132 | 15
Month 3 Primary/Secondary Objectives | 42 (As prespecified, the primary objective included the first 42 Thoracic/Lumbar RF Ablation subjects to complete Month 3.) | 15 (As prespecified, the secondary objective included all Periacetabulum/Iliac Crest/Sacrum RF Ablation subjects.)
Month 6 | 101 | 13
Completed (The objectives are based on Month 3 outcomes (study 'Completed' is Month 12). The study ended when all subjects completed the 6 month visit.) | 51 | 8
Not Completed | 133 | 14

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is based on all subjects treated with RF Ablation.
Groups:
- Total: Total of all reporting groups
Arm/Group | OsteoCool™ RF Ablation in Thoracic/Lumbar Spine | OsteoCool™ RF Ablation in Periacetabulum/Iliac Crest/Sacrum | Total
Number analyzed (Participants) | 184 | 22 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (13.4) | 65.3 (9.4) | 63.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 8 | 113
  Male | 79 | 14 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 150 | 18 | 168
  Canada | 27 | 4 | 31
  France | 6 | 0 | 6
  Germany | 1 | 0 | 1
Wost Pain Score [Mean (Standard Deviation); unit: units on a scale] — Worst pain score (WPS) at the target treatment site in the previous 24 hours was collected using the Brief Pain Inventory (BPI). The WPS is a single question from the BPI (scored from 0-10; 0=NO PAIN and 10=PAIN AS BAD AS YOU CAN IMAGINE). Lower scores indicate less pain.
  units on a scale | 7.8 (1.7) | 7.9 (1.4) | 7.8 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change of Worst Pain Score: Thoracic/Lumbar Spine RF Ablation
Description: Demonstrate an improvement of worst pain score (WPS) at the target treatment site in the previous 24 hours for subjects with metastatic lesions in only the thoracic and/or lumbar vertebral body(ies) as collected using the Brief Pain Inventory (BPI). The WPS is a single question from the BPI (scored from 0-10; 0=NO PAIN and 10=PAIN AS BAD AS YOU CAN IMAGINE). Lower scores indicate less pain.
Time Frame: From Baseline to 3 months post RF ablation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- OsteoCool™ RF Ablation in Thoracic/Lumbar Spine: Subjects with metastatic lesions in only the thoracic and/or lumbar vertebral body(ies).
Arm/Group | OsteoCool™ RF Ablation in Thoracic/Lumbar Spine
Number analyzed (Participants) | 42
units on a scale | -4.1 [-5.2 to -3.1]
Statistical Analysis 1: Comparison: OsteoCool™ RF Ablation in Thoracic/Lumbar Spine; An improvement from baseline to 3 months post radiofrequency ablation in worst pain score will be demonstrated with an outcome which is statistically lower than zero; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Change in Worst Pain Score: Periacetabulum, Iliac Crest, and/or Sacrum RF Ablation
Description: Characterize change in worst pain score (WPS) at the target treatment site in the previous 24 hours for subjects with metastatic lesions in the periacetabulum, iliac crest, and/or sacrum as collected using the Brief Pain Inventory (BPI). Some subjects also had an additional thoracic/lumbar ablation. The WPS is a single question from the BPI (scored from 0-10; 0=NO PAIN and 10=PAIN AS BAD AS YOU CAN IMAGINE). Lower scores indicate less pain.
  The secondary outcome is based on a mutually exclusive cohort of study subjects as compared to the primary outcome.
Time Frame: From Baseline to 3 months post RF ablation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OsteoCool™ RF Ablation in Periacetabulum/Iliac Crest/Sacrum
Number analyzed (Participants) | 15
units on a scale | -4.5 [-6.1 to -2.8]

ADVERSE EVENTS:
Time Frame: From RF Ablation to Month 12.
Description: AE data are based on all available safety data (ie, based on 206 total subjects undergoing RF Ablation including 184 in only the thoracic and/or lumbar vertebral body(ies) and 22 in the periacetabulum, iliac crest, and/or sacrum).
  Device, therapy, and procedure related AEs were considered reportable. Deaths due to underlying malignancy were not considered AE; all deaths were reviewed for causality by a Clinical Events Committee.
Groups:
- Total OsteoCool™ RF Ablation: Subjects underwent a single OsteoCool™ RF Ablation procedure.
  OsteoCool™ RF Ablation: The OsteoCool™ RF Ablation system is indicated in the United States (US), Europe (EUR) and Canada (CAN) for patients with metastatic malignant lesions in a vertebral body, painful metastatic lesions involving bone (in the US, patients with metastatic lesions involving the bone must have failed or were not candidates for standard therapy) and benign bone tumors such as osteoid osteomas.
Arm/Group | Total OsteoCool™ RF Ablation
All-Cause Mortality (participants affected / at risk) | 82/206
Serious Adverse Events (participants affected / at risk) | 3/206
Other Adverse Events (participants affected / at risk) | 0/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total OsteoCool™ RF Ablation (N=206)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participating Institutions may publish the results provided that any such Publication shall be after the multi-center publication is released or presented and shall be provided to Medtronic for review at least 30 days prior to submission or presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT03249584/Prot_SAP_000.pdf